CLINICAL TRIAL: NCT02461134
Title: A Phase 2, Open-label, Single-arm, Intra-subject Dose-escalation Study to Investigate the Biological Activity, Safety, Tolerability, and Pharmacokinetics of Ponesimod in Subjects With Symptomatic Moderate or Severe Chronic GVHD Inadequately Responding to First or Second Line Therapy
Brief Title: Clinical Study to Investigate the Biological Activity, Safety, Tolerability, and Pharmacokinetics of Ponesimod in Subjects With Symptomatic Chronic GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-058C202
Record Dates: First submitted 2015-04-28; First posted 2015-06-03 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Chronic Graft Versus Host Disease
Keywords: GVHD; ponesimod
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ponesimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ponesimod (Experimental): Study treatment consists of 3 consecutive periods: 5 mg ponesimod treatment period (including up-titration), 10 mg treatment period (including up-titration) and a 20 mg treatment period.
  Interventions: Drug: Ponesimod

INTERVENTIONS:
Drug: Ponesimod — Oral film-coated tablets at the doses of 2, 3, 4, 5, 6, 7, 8, 9, 10, and 20 mg. One tablet of ponesimod at any dose will be taken orally once daily.
  Other Names: ACT-128800

SUMMARY:
Chronic graft versus host diseasre (GVHD) is a serious reaction that might occur in a person (the host) who has received cells or organs (graft) from another person because the graft attacks the host's cells. Currently there are no approved therapies for chronic GVHD in the USA, and patients with chroninc GVHD are treated with immunosuppressant drugs. T-lymphocytes (a type of white blood cells) are likely to play a role in the development of chronic GVHD. Due to the capacity of ponesimod to block the traffic of T-lymphocytes, ponesimod may be a new therapeutic approach to treat chroninc GVHD.

The main objective of this study is to assess the effectiveness and safety of several doses of ponesimod in subjects with chronic GVHD who did not respond to standard available treatments.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Symptomatic moderate or severe chronic GVHD patients in need of a change of systemic immunosuppressant (IS) therapy
* Women of child bearing potential must have a negative pregnancy test and use reliable methods of contraception

Exclusion Criteria:

* Clinically significant medical conditions including active or uncontrolled infections, new or recurrent malignancy, serious cardiac, pulmonary, or renal disease, and uncontrolled diabetes.
* Karnofsky Performance Score < 60.
* Immunosuppressant therapies other than allowed background therapy
* Anti-arrhythmic and heart rate lowering drugs.
* Any other circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniele D'Ambrosio, MD, PhD, Study Chair — Actelion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 subjects were screened at 5 different sites. 1 subject was finally recruited into the study. The study was prematurely terminated due to poor recruitment.
Pre-assignment Details: The protocol-defined study population included male and female subjects aged 18 to 70 years with chronic Graft versus Host disease (GVHD). It was planned to recruit 30 subjects.
Groups:
- Ponesimod: It was planned that enrolled subjects receive ponesimod in escalating doses of 5, 10 and 20 mg over the course of the treatment period of 24 weeks in total (4 weeks of 5 mg incl. up-titration, 4 weeks of 10 mg incl. up-titration and 16 weeks of 20 mg).
Period: Overall Study
Arm/Group | Ponesimod
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ponesimod
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Peripheral Absolute Lymphocyte Count From Baseline to Week 4, 8 and 12
Description: The primary pharmacodynamic endpoint assesses intra-subject dose response during the first 12 weeks of treatment.
Time Frame: From baseline to Week 12
Population: Due to the premature termination of the study and consequent lack of meaningful data, no analyses were performed. The statistical analysis plan issued is obsolete, it was not finalized and was therefore not executed.
Arm/Group | Ponesimod
Number analyzed (Participants) | 0

2. Secondary Outcome: Incident Rate of Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: This outcome measure reports the occurrence of adverse events (AEs), and serious adverse events (SAEs) during the treatment period and the follow-up period, and AEs leading to premature discontinuation of study drug. A treatment-emergent AE is any AE temporally associated with the use of study treatment whether or not considered by the investigator as related to study treatment.
Time Frame: From the first study drug intake up to 30 days after last study drug intake (Week 24)
Population: The premature termination of the study led to a consequent lack of meaningful data. As the statistical analysis plan issued was not finalized and was not executed, no statistical analyses were performed. As there was only 1 patient enrolled in the study, the safety events reported occur with 100% frequency.
Measure: Count of Participants; unit: Participants
Arm/Group | Ponesimod
Number analyzed (Participants) | 1
Participants
  Participants with AEs | 1
  Participants with SAEs | 1
  Participants discontinued prematurely study drug | 1

3. Other Pre Specified Outcome: Assessment of a Partial or Complete Overall Response at Week 24
Description: The exploratory efficacy endpoint is based on the 2014 NIH Consensus Development Project response criteria. A complete overall response is defined as a resolution of all reversible manifestations due to chronic GVHD in each organ as defined per NIH Consensus Development Project response criteria. A partial overall response is defined as improvement in a measure for at least one organ without progression in measures for any other organ.
Time Frame: At Week 24
Population: as for outcome 1
Arm/Group | Ponesimod
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study treatment was terminated on Day 81 and the subject was exposed to ponesimod for a total of 81 days (i.e., Day 1 to Day 81). None of the reported adverse events (AEs) were considered by the investigator to be related to the study drug. As there was only 1 patient enrolled in the study, all (S)AEs reported occur with 100% frequency.
Description: All AEs were coded using MedDRA version 19.0. No AEs were reported during the screening period.
Arm/Group | Ponesimod
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponesimod (N=1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Virus infection (Infections and infestations) | 1 (1)
Haematemesis, Parainfluenza (Gastrointestinal disorders) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ponesimod (N=1)
Atrial flutter (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to poor recruitment with 1 subject enrolled. Due to consequent lack of meaningful data, no conclusive analyses could be performed. The statistical analysis plan is obsolete and therefore not applicable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT02461134/Prot_SAP_000.pdf